CLINICAL TRIAL: NCT06334653
Title: Exercise-regulated Organ Crosstalk, Influence of IL-6
Acronym: EVEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helga Ellingsgaard (Other)
Responsible Party: Sponsor-Investigator, Helga Ellingsgaard, Principle Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-23069670
Record Dates: First submitted 2024-03-13; First posted 2024-03-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-04

CONDITIONS: Healthy Volunteers Only; Energy Metabolism
Keywords: tocilizumab; exercise; IL-6; extracellular vesicles; energy; muscle; liver; brain
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Saline infusion
  Interventions: Other: exercise
- Tocilizumab (Experimental): IL-6 receptor antibody infusion (8 mg/kg body weight, max 800 mg)
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — acute exercise bout

SUMMARY:
Overall the study investigates organ crosstalk during exercise. More specifically, the study investigates the role of IL-6 in regulating glucose, fatty acid, and amino acid kinetics at whole body level and in skeletal muscle, liver, and brain. Furthermore, the study investigates the uptake and release of extracellular vesicles in skeletal muscle, liver, and brain in reponse to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 18 years
* Maximum age: 45 years
* Minimum BMI: 18
* Maximum BMI: 25
* Sex: Male
* Healthy (based on screening)
* Stable body weight for 6 months
* VO2max (mL/kg/min) ≥ 50

Exclusion Criteria:

* Smoking
* Thyroid disease
* Heart disease
* Inflammatory diseases
* Current infection
* Liver disease (transaminases more than 2x upper normal range)
* Kidney disease (creatinine more than1.5 mg/dl)
* Known immunosuppressive disease
* Corticosteroid use
* Regular NSAID or paracetamol usage
* Aspirin use more than 100 mg/d
* History of carcinoma
* History of tuberculosis
* Anemia (hematocrit less than 33%)
* WBC less than 1 x 10^3
* Platelets less than 100 x 10^3
* Bleeding disorders
* Obstructive pulmonary disease
* Femoral hernia
* Vascular prosthesis
* Vascular thrombosis
* Previous nerve damage
* Many previous femoral catheter installations

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Whole body substrate kinetics. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing rates of appearances (Ra) and disappearances (Rd) of glucose, glycerol, palmitate, amino acids between placebo and IL-6R ab at rest, during exercise, and recovery.
Tissue specific utilization and production of substrates. | Comparisons between study arms are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing, between placebo and IL-6Rab, by measuring in plasma, the Ra and Rd of substrates in muscle, liver, and brain at rest, during exercise, and recovery using the non-steady-state equations of Steele adapted for stable isotopes.
IL-6 regulation of protein synthesis and degradation. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing differences in protein synthesis and degradation rates between placebo and IL-6Rab at rest, during exercise, and during recovery from exercise.
Number of EVs from muscle, liver, and brain. | Comparisons between placebo and IL-6R ab are done before exercise (time points 255 and 270 minutes).
  Comparing the number of EVs deriving from skeletal muscle, liver, and brain.
Size of EVs from muscle, liver, and brain. | Comparisons between placebo and IL-6R ab are done before exercise (time points 255 and 270 minutes).
  Comparing EV size deriving from skeletal muscle, liver, and brain.
EVs from muscle, liver, and brain. | Comparisons between placebo and IL-6R ab are done before exercise (time points 255 and 270 minutes).
  Comparing the content of EVs deriving from skeletal muscle, liver, and brain.
Influence of exercise on EV number. | Comparisons between placebo and IL-6R ab are done throughout a 1-hour exercise bout (time points 285, 300, 315, and 330 minutes).
  Comparing the number of EVs deriving from skeletal muscle, liver, and brain in response to exercise.
Influence of exercise on EV size | Comparisons between placebo and IL-6R ab are done throughout a 1-hour exercise bout (time points 285, 300, 315, and 330 minutes).
  Comparing EV size deriving from skeletal muscle, liver, and brain in response to exercise.
Influence of exercise on EV content. | Comparisons between placebo and IL-6R ab are done throughout a 1-hour exercise bout (time points 285, 300, 315, and 330 minutes).
  Comparing the content of EVs deriving from skeletal muscle, liver, and brain in response to exercise.
Tissue specific proteomic content of EVs. | Comparisons between placebo and IL-6R ab are done at the end of a 1-hour exercise bout (330 minutes).
  Comparing differences in proteomic content of EVs from skeletal muscle, liver, and brain in response to exercise.

SECONDARY OUTCOMES:
Lactate. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Differences in plasma lactate from skeletal muscle, liver, and brain comparing placebo and IL-6R ab.
Pyruvate. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Differences in plasma pyruvate from skeletal muscle, liver, and brain comparing placebo and IL-6R ab.
Keto acids. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Differences in plasma keto acids from skeletal muscle, liver, and brain comparing placebo and IL-6R ab.
Ketone bodies. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Differences in plasma ketone bodies from skeletal muscle, liver, and brain comparing placebo and IL-6R ab.
Influence of IL-6 on fatty acid oxidation rates. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing, between placebo and IL-6R ab, differences in fatty acid, e.g. palmitate oxidation rates, at whole body level and in skeletal muscle, liver, and brain.
Influence of IL-6 on insulin. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing differences in plasma insulin concentrations between placebo and IL-6R ab.
Influence of IL-6 on glucagon. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing differences plasma glucagon concentrations between placebo and IL-6R ab.
Influence of IL-6 on epinephrine. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing differences in plasma epinephrine concentrations between placebo and IL-6R ab.
Influence of IL-6 on norepinephrine. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing differences in plasma norepinephrine concentrations between placebo and IL-6R ab.
IL-6 levels. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Comparing differences in plasma IL-6 concentrations between placebo and IL-6R ab.
Influence of IL-6 on substrate usage. | Comparisons between placebo and IL-6R ab are done at rest (time points 255 and 270 minutes), during exercise (time points 285, 300, 315, and 330 minutes) and during recovery from exercise (time points 345, 360, and 390 minutes).
  Differences in respiratory exchange ratio comparing placebo and IL-6R ab.
Influence of IL-6 on perceived exertion. | Comparisons between placebo and IL-6R ab are done during exercise (time points 285, 300, 315, and 330 minutes).
  Differences in rate of perceived exertion during exercise comparing placebo and IL-6R ab.

CONTACTS AND LOCATIONS:
Overall Officials: Helga Ellingsgaard, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No